CLINICAL TRIAL: NCT04516642
Title: Swiss Frailty Network and Repository
Acronym: SFNR
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Zurich (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other); University Department of Geriatric Medicine FELIX PLATTER (Other); University Hospital, Geneva (Other); University of Lausanne Hospitals (Other)
Responsible Party: Sponsor
Other Study IDs: SPHN Project-ID 2017DRI02
Record Dates: First submitted 2020-07-21; First posted 2020-08-18 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Weight Loss; Fatigue; Physical Frailty; Weakness, Muscle
Keywords: Frailty; Frailty-Index
MeSH Terms: conditions — Weight Loss; Fatigue; Muscle Weakness; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Physical frailty is an age-related medical syndrome defined by a decline in multiple body systems, thus causing increased vulnerability, even in the face of minor stressors (1) It has been linked to multiple negative health outcomes, including extended length of stay in acute care due to complications, hospital re-admissions, and mortality among older patients. About 10-30% of community-dwelling seniors are considered frail(2) with an additional 40% being at risk for the condition (pre-frailty). By 2030, the number of older adults with frailty is expected to at least double, in parallel to the projected growth of the older segment of the population. Frail seniors consume 3-times more health care resources then their robust counterparts. Thus, the health economic impact of frailty is expected to be enormous and a call to action has been posed. Big data in healthcare provides important opportunities for the identification of frailty among the growing number of older patients. This is relevant as frailty is considered a better predictor of adverse outcomes than chronological age alone. Therefore, several medical specialties have started to assess frailty in cancer patients, heart surgery candidates and potential organ transplant recipients.

DETAILED DESCRIPTION:
The Swiss Frailty Network and Repository is a Swiss Personalized Health Network (SPHN) driver project. The investigators aim to promote the sustainable implementation of a frailty data network for research and clinical purposes in strong partnership between all Swiss geriatric academic centers.

One of the five main goals of this project is to validate an electronic frailty index (eFI) as a screening tool against a clinical frailty instrument (cFI) (validation study) and the investigation of the correlation of the two instruments with the important endpoints in-hospital mortality and length of stay in hospital (association study) is at the core of the project. For the validation study (4), the investigators will include patients 65 and older admitted to acute geriatric care at all partnering sites, where both, the cFI and the eFI is collected. For the validation study (4), the investigators will include only patients with written project informed consent and consent for subsequent use of the project data (the investigators will also ask for general consent whenever possible. For the correlation study (5) regarding the cFI and the 2 outcomes. The same requirements apply as for the validation study (4). For the association study (5) regarding the eFI screening tool, the investigators will utilize data from all patients age 65 and older admitted to acute care at all partnering sites. For the eFI, the investigators will only include participants with available written general consent for further use of routinely collected health data, or established permission for use in exceptional cases by an ethics committee (HRA Art. 34).

Due to time constraints and great complexity of the local integration of the clinical frailty instrument (cFI) as a reference measure at the five different clinic information systems, the investigators will only integrate the cFI into the primary system at University Hospital Zurich (USZ) during the three-year duration of the project. At all other partner sites, an electronic case report form in REDCap will be in place for data entry of the cFI assessment.

In summary, the investigators will categorize the collection of data for the clinical Frailty Instrument (cFI) and the electronic Frailty Index (eFI) screening tool in geriatric inpatients 65 years and older (validation study plus correlation study) at all sites as a category A research project (not a clinical trial) with only minimal risks at all partner sites and the collection of the eFI screening tool in all other acute care patients 65 years and older as a further use of non-genetic personal health data in patients where a general consent is available.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 65 and older
* Admission as inpatients to acute care at any partnering university hospital (eFI - subgroup)
* Admission as inpatients to acute geriatric care (cFI - subgroup)
* Patients or proxies need to provide a written informed consent (geriatric patients (cFI and eFI): project consent; non-geriatric patients ((eFI): general consent)

Exclusion Criteria:

* Documented objection of participating in the project and/or subsequent use of personal health data
* Not fluent in local language (i.e. German, French)
* Patient is uncooperative or presence of inability to perform functional tests due to severe cognitive and/or physical impairment/acute medical illness

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Hospitalized patients age 65 and older from all 5 university hospitals in Switzerland (Basel, Bern, Geneva, Lausanne and Zurich)
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Positive and negative predictive value of the eFI | year 2-3
  Validation Study
sensitivity and specificity of the eFI | year 2-3
  Validation Study
The correlation between the cFI and the eFI with length of stay and in-hospital mortality | year 2-3
  Correlation Study

CONTACTS AND LOCATIONS:
Overall Officials: Heike Bischoff-Ferrari, MD, DrPH, Principal Investigator — University of Zurich
Locations (1):
- Dept. of Geriatrics and Aging Research, University of Zurich / Geriatric Clinic University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
The investigators will categorize the collection of the data for the clinical Frailty Instrument (cFI) and the electronic Frailty Index (eFI) screening tool in geriatric inpatients 65 years and older (validation study plus association study) at all sites as a category A research project (not a clinical trial) with only minimal risks at all partner sites and the collection of the eFI screening tool in all other acute care patients 65 years and older as a further use of non-genetic personal health data in patients where a general consent is available.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: In order to ensure the same quality and standards between all 5 sites, data analysis, instructor training and project documents will be shared.
Access Criteria: Personnel of the departments of geriatrics involved in our SFNR project at each center (Basel, USB and Felix Platter Spital], Bern [INSEL and Spital Tiefenau], Geneva [HUG], Lausanne [CHUV] and Zurich [USZ]) and collaborating Research Data Warehouses of the aforementioned locations are entitled to pass on the personal data. In addition, the investigators entitle the responsible physicians of all involved acute care wards (i.e. general internal medicine and medical subspecialties, general surgery and surgical subspecialties, oncology, haematology, intensive care, neurology, dermatology, rheumatology, ophthalmology, emergency medicine, gynaecology, ENT/ORL, urology) at the partnering hospitals to pass on the routinely collected data for the eFI variables. A data transfer agreement will be established among all co-investigators before data transfer begins.

REFERENCES:
- [Derived] Gagesch M, Edler K, Chocano-Bedoya PO, Abderhalden LA, Seematter-Bagnoud L, Meyer T, Bertschi D, Zekry D, Bula CJ, Gold G, Kressig RW, Stuck AE, Bischoff-Ferrari HA. Swiss Frailty Network and Repository: protocol of a Swiss Personalized Health Network's driver project observational study. BMJ Open. 2021 Jul 14;11(7):e047429. doi: 10.1136/bmjopen-2020-047429. PMID 34261684